CLINICAL TRIAL: NCT05852093
Title: Clinical Study on the Effect of Tizanidine on the Function and Pain of Patients After Shoulder Arthroscopy
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, YangGuang, Deputy chief doctor, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 研2023-0251
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug: Celecoxib+Buprenorphine Transdermal Patch (Active Comparator)
  Interventions: Drug: Celecoxib+Buprenorphine Transdermal Patch
- Drug: Celecoxib+Buprenorphine Transdermal Patch+Tizanidine (Experimental)
  Interventions: Drug: Celecoxib+Buprenorphine Transdermal Patch+Tizanidine

INTERVENTIONS:
Drug: Celecoxib+Buprenorphine Transdermal Patch — NSAIDs+narcotic analgesics
  Arms: Drug: Celecoxib+Buprenorphine Transdermal Patch
Drug: Celecoxib+Buprenorphine Transdermal Patch+Tizanidine — NSAIDs+narcotic analgesics+Skeletal Muscle Relaxant
  Arms: Drug: Celecoxib+Buprenorphine Transdermal Patch+Tizanidine

SUMMARY:
The perspective, randomized controlled trial is to investigate and evaluate the effect of Tizanidine on the function and pain of patients with rotator cuff tear after shoulder arthroscopy;

ELIGIBILITY:
Inclusion Criteria:

1 Patients who were diagnosed as supraspinatus tendon and infraspinatus tendon tear and underwent shoulder arthroscopic surgery in the Second Affiliated Hospital of Zhejiang University; 2 Age 20~70 years old; 3 Those with a long medical history, and symptoms such as shoulder joint pain and weakness in a short period of time are obviously aggravated; 4. After 3 months of medication and physical therapy, the symptoms and functions have not improved significantly; 5 Volunteer to participate in this study, and the person and his/her family members have given informed consent to the content of this study and signed the consent form

Exclusion Criteria:

1. Patients with simple frozen shoulder;
2. Patients with shoulder joint tuberculosis, gout, tumor, rheumatoid disease or infectious disease; 3. There are other joint pain factors before operation;

4 Patients with subscapularis tendon tear, long head tendinopathy requiring surgical treatment, and severe shoulder synovitis were found during the operation; 5 Patients with upper limb nerve injury, shoulder fracture, bone defect or severe osteoporosis; 6. Patients with serious organ or hematopoietic system and other primary diseases; 7. Those who are allergic to the drugs used in this study; 8 Women who are breast-feeding, pregnant or preparing to become pregnant; 9 Patients with language and communication disorders, mental history, cognitive dysfunction, etc. who cannot cooperate with the completion of nursing intervention and research, and cannot complete the questionnaire required for this study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index；PSQI | From Week 0 (baseline) to Week24

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons Score; ASES | From Week 0 (baseline) to Week24
UCLA score; UCLA | From Week 0 (baseline) to Week24
Visual Analogu Scale; VAS | From Week 0 (baseline) to Week24
Oxford Shoulder Score; OSS | From Week 0 (baseline) to Week24

IPD SHARING:
Plan to Share IPD: Yes